CLINICAL TRIAL: NCT01865552
Title: A Randomised, Single-blind, Three-part, Two-period, Two-sequence, Single-dose, Cross-over Study to Compare the Pharmacokinetics, Safety, Tolerability and Immunogenicity of Three Formulations of Etanercept (SB4, EU Sourced Enbrel® and US Sourced Enbrel®) in Healthy Male Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability and Immunogenicity Study of SB4 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SB4-G11-NHV; 2012-004371-39 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- SB4 and EU sourced Enbrel in Part A (Experimental): SB4 followed by EU sourced Enbrel
  Interventions: Biological: SB4; Biological: EU sourced Enbrel
- EU sourced Enbrel and SB4 in Part A (Experimental): EU sourced Enbrel followed by SB4
  Interventions: Biological: SB4; Biological: EU sourced Enbrel
- SB4 and US sourced Enbrel in Part B (Experimental): SB4 followed by US sourced Enbrel
  Interventions: Biological: SB4; Biological: US sourced Enbrel
- US sourced Enbrel and SB4 in Part B (Experimental): US sourced Enbrel followed by SB4
  Interventions: Biological: SB4; Biological: US sourced Enbrel
- EU and US sourced Enbrel in Part C (Other): EU sourced Enbrel followed by US sourced Enbrel
  Interventions: Biological: EU sourced Enbrel; Biological: US sourced Enbrel
- US and EU sourced Enbrel in Part C (Other): US sourced Enbrel followed by EU sourced Enbrel
  Interventions: Biological: EU sourced Enbrel; Biological: US sourced Enbrel

INTERVENTIONS:
Biological: SB4 — SC administration
  Arms: EU sourced Enbrel and SB4 in Part A; SB4 and EU sourced Enbrel in Part A; SB4 and US sourced Enbrel in Part B; US sourced Enbrel and SB4 in Part B
Biological: EU sourced Enbrel — SC administration
  Arms: EU and US sourced Enbrel in Part C; EU sourced Enbrel and SB4 in Part A; SB4 and EU sourced Enbrel in Part A; US and EU sourced Enbrel in Part C
Biological: US sourced Enbrel — SC administration
  Arms: EU and US sourced Enbrel in Part C; SB4 and US sourced Enbrel in Part B; US and EU sourced Enbrel in Part C; US sourced Enbrel and SB4 in Part B

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety and immunogenicity of SB4 and Enbrel (EU sourced Enbrel and US sourced Enbrel) in healthy male subjects.

DETAILED DESCRIPTION:
* Part A: Comparison between SB4 and EU sourced Enbrel
* Part B: Comparison between SB4 and US sourced Enbrel
* Part C: Comparison between EU sourced Enbrel and US sourced Enbrel

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Have a body weight between 60 and 94.9 kg and a body mass index between 20.0 and 29.9 kg/m², inclusive.

Exclusion Criteria:

* history and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to any components of the test and reference IP formulation or comparable drugs.
* active or latent Tuberculosis or who have a history of TB.
* history of invasive systemic fungal infections or other opportunistic infections
* systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
* serious infection associated with hospitalisation and/or which required intravenous antibiotics
* history of and/or current cardiac disease
* have received live vaccine(s) within 30 days prior to Screening or who will require live vaccine(s) between Screening and the final study visit.
* Intake medication with a half-life > 24 h within 1 month or 10 half-lives of the medication prior to the first administration of IP.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, M.D., Ph.D., Principal Investigator — Parexel
Locations (1):
- Parexel International GmbH, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- SB4 and EU Sourced Enbrel in Part A: SB4 (Period 1) followed by EU sourced Enbrel (Period 2)
  SB4: SC administration
  EU sourced Enbrel: SC administration
- EU Sourced Enbrel and SB4 in Part A: EU sourced Enbrel (Period 1) followed by SB4 (Period 2)
  SB4: SC administration
  EU sourced Enbrel: SC administration
- SB4 and US Sourced Enbrel in Part B: SB4 (Period 1) followed by US sourced Enbrel (Period 2)
  SB4: SC administration
  US sourced Enbrel: SC administration
- US Sourced Enbrel and SB4 in Part B: US sourced Enbrel (Period 1) followed by SB4 (Period 2)
  SB4: SC administration
  US sourced Enbrel: SC administration
- EU and US Sourced Enbrel in Part C: EU sourced Enbrel (Period 1) followed by US sourced Enbrel (Period 2)
  EU sourced Enbrel: SC administration
  US sourced Enbrel: SC administration
- US and EU Sourced Enbrel in Part C: US sourced Enbrel (Period 1) followed by EU sourced Enbrel (Period 2)
  EU sourced Enbrel: SC administration
  US sourced Enbrel: SC administration
Period: Period 1
Arm/Group | SB4 and EU Sourced Enbrel in Part A | EU Sourced Enbrel and SB4 in Part A | SB4 and US Sourced Enbrel in Part B | US Sourced Enbrel and SB4 in Part B | EU and US Sourced Enbrel in Part C | US and EU Sourced Enbrel in Part C
Started | 23 | 23 | 23 | 23 | 23 | 23
Discontinued From Period 1 | 1 | 0 | 0 | 1 | 3 | 1
Completed | 22 | 23 | 23 | 22 | 20 | 22
Not Completed | 1 | 0 | 0 | 1 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Pathological lab | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | SB4 and EU Sourced Enbrel in Part A | EU Sourced Enbrel and SB4 in Part A | SB4 and US Sourced Enbrel in Part B | US Sourced Enbrel and SB4 in Part B | EU and US Sourced Enbrel in Part C | US and EU Sourced Enbrel in Part C
Started | 22 | 23 | 23 | 22 | 20 | 22
Completed | 22 | 23 | 23 | 22 | 20 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB4 and EU Sourced Enbrel in Part A | EU Sourced Enbrel and SB4 in Part A | SB4 and US Sourced Enbrel in Part B | US Sourced Enbrel and SB4 in Part B | EU and US Sourced Enbrel in Part C | US and EU Sourced Enbrel in Part C | Total
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9.4) | 41 (10.9) | 38 (9.7) | 43 (8.9) | 40 (10.5) | 41 (9.4) | 40 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 23 | 23 | 23 | 23 | 23 | 23 | 138

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: pre-dose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312 and 480 h post-dose
Time Frame: 0 to 480 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: µg·h/mL
Groups:
- SB4 in Part A; SB4 in Part B: SB4: SC administration
- EU Sourced Enbrel in Part A; EU Sourced Enbrel in Part C: EU sourced Enbrel: SC administration
- US Sourced Enbrel in Part B; US Sourced Enbrel in Part C: US sourced Enbrel: SC administration
Arm/Group | SB4 in Part A | EU Sourced Enbrel in Part A | SB4 in Part B | US Sourced Enbrel in Part B | EU Sourced Enbrel in Part C | US Sourced Enbrel in Part C
Number analyzed (Participants) | 42 | 42 | 44 | 44 | 42 | 42
µg·h/mL | 769.069 (243.9039) | 771.680 (226.2874) | 834.680 (242.7652) | 810.054 (195.9770) | 790.110 (274.2535) | 768.228 (238.1251)

2. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: pre-dose (0 h) and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312 and 480 h post-dose.
Time Frame: 0 to 480 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | SB4 in Part A | EU Sourced Enbrel in Part A | SB4 in Part B | US Sourced Enbrel in Part B | EU Sourced Enbrel in Part C | US Sourced Enbrel in Part C
Number analyzed (Participants) | 42 | 42 | 44 | 44 | 42 | 42
μg/mL | 3.607 (1.4298) | 3.435 (1.2390) | 3.869 (1.3251) | 3.613 (1.0252) | 3.720 (1.5444) | 3.575 (1.4833)

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: pre-dose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312 and 480 h post-dose
Time Frame: 0 to 480 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: µg·h/mL
Arm/Group | SB4 in Part A | EU Sourced Enbrel in Part A | SB4 in Part B | US Sourced Enbrel in Part B | EU Sourced Enbrel in Part C | US Sourced Enbrel in Part C
Number analyzed (Participants) | 42 | 42 | 44 | 44 | 42 | 42
µg·h/mL | 728.169 (234.7621) | 734.015 (220.2722) | 788.773 (232.4636) | 765.187 (184.5046) | 752.277 (259.2088) | 727.820 (229.8597)

4. Secondary Outcome: Time to Cmax (Tmax)
Description: pre-dose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312 and 480 h post-dose
Time Frame: 0 to 480 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SB4 in Part A | EU Sourced Enbrel in Part A | SB4 in Part B | US Sourced Enbrel in Part B | EU Sourced Enbrel in Part C | US Sourced Enbrel in Part C
Number analyzed (Participants) | 42 | 42 | 44 | 44 | 42 | 42
h | 75.198 (29.1358) | 71.711 (24.7538) | 75.263 (30.8374) | 70.385 (22.4972) | 70.276 (30.3826) | 71.150 (29.7904)

ADVERSE EVENTS:
Time Frame: 7 weeks (49 days) after first dose administration of SB4, EU sourced Enbrel, or US sourced Enbrel
Arm/Group | SB4 in Part A | EU Sourced Enbrel in Part A | SB4 in Part B | US Sourced Enbrel in Part B | EU Sourced Enbrel in Part C | US Sourced Enbrel in Part C
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46 | 0/46 | 0/46 | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46 | 0/46 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 18/46 | 16/46 | 23/46 | 20/46 | 17/46 | 14/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB4 in Part A (N=46) | EU Sourced Enbrel in Part A (N=46) | SB4 in Part B (N=46) | US Sourced Enbrel in Part B (N=46) | EU Sourced Enbrel in Part C (N=46) | US Sourced Enbrel in Part C (N=46)
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 0
Lip erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 2 | 3 | 3 | 3 | 1 | 3
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 2 | 2 | 1
Rhinitis (Infections and infestations) | 2 | 2 | 1 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 3 | 4 | 4 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 2 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes